CLINICAL TRIAL: NCT02607787
Title: The Feasibility and Effects of a Home-based Walking and Strengthening Intervention on Physiological, Biochemical and Psychological Outcomes in Colo-rectal Cancer Survivors
Brief Title: EXercise And Colo-Rectal Cancer Trial
Acronym: EXACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14/0061 (EXACT Study); 14127JG-SS (Other: HSC Trust UK); 14/NI/1048 (Other: ORECNI)
Record Dates: First submitted 2015-07-08; First posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Colo-rectal Cancer
Keywords: Exercise Rehabilitation
MeSH Terms: conditions — Colonic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group (Experimental): As well as usual care, this group receive a behavioural change session and intervention information regarding the exercise programme. The home-based walking and strengthening intervention is individually tailored for each participant. They receive a booklet, diary and pedometer to guide them as well as weekly phone calls for 12 weeks to monitor their progress.
  Interventions: Behavioral: Exercise
- Control Group (Other): This group attends and participates in the same assessment outcomes as the intervention group and receives usual care for the duration of the study. However they are not given any exercise instructions and do not receive the intervention information until their final assessment at week 24. They are aware of their group allocation throughout the duration of the study.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Exercise — The exercise programme aims to gradually increase participants physical activity levels so that they start achieving the recommended levels of at least 150 minutes moderate intensity aerobic activity per week and strengthening exercise for all major muscle groups at least twice per week.
  Arms: Exercise Group
Other: Control — The control group will receive usual care whilst attending for the same 4 visits as the intervention group and have the same outcome measures tested. They will however receive the intervention information on their last visit.
  Arms: Control Group

SUMMARY:
The aim of this study is to assess the feasibility and effectiveness of a home-based walking and strengthening intervention on physiological, biochemical and psychological outcomes in colo-rectal cancer survivors.

The intervention consists of a 12-week home-based walking and strengthening programme for colo-rectal cancer survivors post any anti-cancer treatment. It aims to gradually increase participants physical activity levels so that they start achieving the recommended levels of at least 150 minutes moderate intensity aerobic activity per week and strengthening exercise for all major muscle groups at least twice per week.

As well as usual care, the intervention group will receive weekly telephone calls and a behaviour change interview at baseline. Participants will be recruited from the Cancer Centre at the Belfast City Hospital. Assessments will be taken at baseline (0 weeks), post intervention (12 weeks) and also at a 3-month follow-up (24 weeks). The control group will receive the same assessments at the same time-points however they will continue to receive usual care with the intervention information (including pedometer, exercise booklet, diary and behavioural change interview) being given at the 3-month follow-up appointment.

DETAILED DESCRIPTION:
The number of people living with and beyond cancer is ever increasing and now more than ever there is a need to facilitate the appropriate rehabilitation of these patients. Exercise interventions and increased physical activity have been well documented in their ability to improve multiple aspects of health in cancer survivors; including quality of life, fatigue as well as all-cause and cancer-specific mortality. Whilst the main outcome from this study will be its feasibility, the novel aspect is the analysis of biological markers in the blood. Although there is much evidence on the benefits of exercise for colo-rectal cancer survivors, the biological mechanisms underlying its effects in this population are still elusive. Therefore this intervention was designed to investigate the feasibility and effectiveness of a home-based walking and strengthening programme on physiological, biochemical and psychological outcomes in colo-rectal cancer survivors.

Participants are first approached by their surgeon/oncologist and assessed for their eligibility. If they are deemed eligible they are then referred to the researcher in the waiting room to be given more information about the study. If interested, they receive the participant information sheet and consent forms to take home for a period of at least 24 hours, after which the researcher calls to confirm their interest. Visit 1 is then scheduled in order for the participant to sign the consent forms and receive the 'ActiGraph' accelerometer which they wear for 7 consecutive days in order to measure their baseline physical activity levels. With permission, the patients GP will be advised by letter that the patient is commencing the study.

After the seven days the participant attends the Northern Ireland Clinical Research Facility at the Belfast City Hospital for the first assessment session. The outcome measures assessed include analysis on feasibility, quality of life, fatigue, biological markers, anthropometry, strength, cardiovascular endurance and physical activity levels. The intervention group then receive the behaviour change counselling session along with the exercise booklet, diary and pedometer. Weekly phone calls are made to intervention participants for 12 weeks to monitor their progress. The control group receives usual care without weekly phone calls. On week 11 both groups are posted their accelerometer to record activity levels and then attend the City Hospital to repeat all assessments. Both groups are not contacted again until week 23 when they are posted the accelerometer for the final time and their follow-up assessments are complete. It is at this assessment session that the control group receive the behaviour change session and intervention materials.

After each assessment day, blood samples are transported via a specifically designed fridge, to the Ulster University campus to be stored at -80 degrees Celsius for future analysis. All other study information such as questionnaires and collected data are stored as per University protocol in storage containers in a designated locked room on campus.

ELIGIBILITY:
Inclusion Criteria:

* Dukes A-C colo-rectal cancer patients at least 6 weeks post any-type anti-cancer treatment, as identified by the colo-rectal oncologic and surgical teams at the Cancer Centre, Belfast City Hospital, Belfast Health and Social Care Trust.
* Males and females.
* Over eighteen years of age.
* Physically able to undertake the intervention as described within the HBWS programme by Donnelly and colleagues (2010).
* Ambulatory and without use of a walking aid.

Exclusion Criteria:

* Still undergoing and/or scheduled for further anti-cancer treatment.
* Any presence of cognitive impairment.
* Known co-morbidities which would severely impact upon physical functioning or nutritional status such as poorly controlled diabetes, heart failure, unstable angina, degenerative neuromuscular disease, inborn errors of metabolism, mental health disorder or substance abuse.
* Already meeting the current recommended physical activity guidelines (Schmitz, et al. 2010).
* Unable to understand and communicate in written and oral English and over the phone sufficiently well enough to undertake the self-management programme and weekly telephone review.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 24 months
  The feasibility of the trial will be characterized by recording such things as; the number of eligible patients, the follow-up rates, response rates to questionnaires and adherence/compliance rates.

SECONDARY OUTCOMES:
Physical activity | For 7 days at three different times; baseline, week 11 and week 23.
  The participants will wear an 'ActiGraph' accelerometer around their waist for 7 consecutive days in order to calculate their activity levels.This will be measured by analyzing the minutes spent in moderate/vigorous/sedentary behaviour.
Cardiovascular Endurance | Week 0, 12 and 24
  Participants walk between two cones 30 metres apart for six minutes. The cones are in a closed off corridor in the hospital with no obstructions. This is measured in meters covered in the 6 minutes.
Lower limb strength | Week 0, 12 and 24
  The 30 second sit-to-stand test requires the participants to sit down and stand up from a chair as many times as they can in 30 seconds. The outcome is the number of repetitions completed.
Quality of life | Week 0, 12 and 24
  Various validated questionnaires will be given to assess quality of life and fatigue; Positive and Negative Affect Schedule (PANAS), EQ-5D-3L questionnaire, FACT-C and FACT-F.
Demographics | Week 0, 12 and 24
  A specially designed demographics questionnaire to gain an insight into the participant characteristics. Outcomes measured will be; age/ethnicity/employment status/marital status.
Height | Week 0, 12 and 24
  Height will be measured in metres/cm.
Venous blood sample | Week 0, 12 and 24
  A 34ml venous blood sample will be taken to measure various markers.
Weight | Week 0, 12 and 24
  Weight will be measured in kg.
Hip and waist circumference | Week 0, 12 and 24
  Measured using a measuring tape in cm.
Capillary blood sample | Week 0, 12 and 24
  Finger prick test performed to measure metabolism related markers.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Gracey, PhD, Principal Investigator — Ulster University
Locations (1):
- Belfast City Hospital, Belfast, Antrim, United Kingdom